CLINICAL TRIAL: NCT02637622
Title: Advancing Stated-preference Methods for Measuring the Preferences of Patients With Type II Diabetes
Brief Title: Measuring the Preferences of Patients With Type II Diabetes Using Best-worst Scaling and Discrete Choice Experiment
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI 90056532 PF
Record Dates: First submitted 2015-11-18; First posted 2015-12-22 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Type II Diabetes
Keywords: conjoint analysis; stated-preference methods; patient centered outcome research (PCOR); community-based participatory research (CBPR); patient preference; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Preference; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Best-Worst Scaling (Case 2): Preference measured by best-worst scaling (case 2)
  Interventions: Other: Best-Worst Scaling (Case 2)
- Discrete Choice Experiment: Preference measured by discrete choice experiment
  Interventions: Other: Discrete Choice Experiment

INTERVENTIONS:
Other: Best-Worst Scaling (Case 2) — Respondents receive questions asking them to choose the best and worst features of a hypothetical medication.
  Groups: Best-Worst Scaling (Case 2)
Other: Discrete Choice Experiment — Respondents receive questions asking them to choose the medication they prefer between a pair of hypothetical medications.
  Groups: Discrete Choice Experiment

SUMMARY:
In 2012, the FDA Center for Devices and Radiological Health (CDRH) issued guidance to clarify the principal benefit-risk factors FDA considers during the reviews for premarket approval applications and de novo classification requests. In addition to a detailed description of benefits and risks, CDRH listed "patient tolerance for risk and perspective on benefit" as a factor that CDRH may consider in regulatory reviews. It underlined the need for developing methods to measure patient preference and incorporate it into regulatory decision-making. The purpose of this study is to advance methods for patient and community engagement in patient-centered outcome research (PCOR) and has three objectives.

First, demonstrate good practices for patient and community involvement in PCOR projects by applying principles of community-based participatory research (CBPR).

Second, address methodological gaps pertaining to the use of stated-preference methods in studying preferences in PCOR. These include identifying the best methods for designing a preference study and strategies for analyzing variation in preferences. The investigators also seek to assess the relevance of stated-preference methods to patients and stakeholders using both qualitative and quantitative methods.

Third, demonstrate good practices for applying stated-preference methods by studying the preferences of patients with type II diabetes. While type II diabetes provides an important case study, this research will advance approaches and methods that will be broadly generalizable to other diseases, and to diverse patient and stakeholder groups.

Clinical Significance:

This project will illustrate and advance methods for assessing the values of patients and stakeholders. It will demonstrate how CBPR methods apply to PCOR studies and the value of stated-preference methods in measuring the preferences of patients and stakeholders and directing health care.

DETAILED DESCRIPTION:
This study will apply the principles of CBPR to involve patients and stakeholders associated with a local community board and a national diabetes advisory board in key decisions in the project. During year 1, the investigators will utilize mixed methods to develop, pretest, and pilot the survey instruments to assess the preferences of patients with type II diabetes. In year 2, the investigators plan further engagement to finalize the survey instruments, and will implement a nationally representative, racially/ethnically diverse sample of patients with type II diabetes. Based on further consultation, the investigators will conduct statistical analysis, including stratified analyses and segmentation of patients with similar preferences. In year 3, mixed methods will be applied to assess beliefs of patients and other consumers about the relevance of this work and its generalizability to other PCOR topics. Finally, lay language reports will be developed to highlight patient and stakeholder engagement and the application of stated-preference methods to the study of the preferences of patients with type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the GfK's KnowledgePanel
* Self-reported Type II diabetes diagnosis

Exclusion Criteria:

* Does not have Type II diabetes diagnosis
* Unable to communicate in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type II diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1103 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bridges, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The survey was conducted through GfK KnowledgePanel. Eligible members were invited by email to participate in the survey. All participants were required to be 18 years or older with self-reported physician-diagnosed type 2 diabetes and able to read English or Spanish. African Americans and Latinos were oversampled.
Pre-assignment Details: 638 respondents (34%) did not respond to the survey and 139 people among those who responded (11%) were excluded based on the screening questions.
Period: Overall Study
Arm/Group | Best-Worst Scaling (Case 2) | Discrete Choice Experiment
Started | 551 | 552
Completed | 551 | 552
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Respondents who completed the survey.
Groups:
- Best-Worst Scaling (BWS) (Case 2): Preference measured by best-worst scaling (case 2)
  Best-Worst Scaling (Case 2): Respondents receive questions asking them to choose the best and worst features of a hypothetical medication.
- Discrete Choice Experiment (DCE): Preference measured by discrete choice experiment
  Discrete Choice Experiment: Respondents receive questions asking them to choose the medication they prefer between a pair of hypothetical medications.
- Total: Total of all reporting groups
Arm/Group | Best-Worst Scaling (BWS) (Case 2) | Discrete Choice Experiment (DCE) | Total
Number analyzed (Participants) | 551 | 552 | 1103
Age, Continuous [Mean (Full Range); unit: years] | 62.55 [25 to 89] | 61.30 [24 to 91] | 61.93 [24 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 279 | 553
  Male | 277 | 273 | 550
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 286 | 289 | 575
  Black, Non-Hispanic | 128 | 126 | 254
  Other, Non-Hispanic | 20 | 18 | 38
  Hispanic | 117 | 119 | 236
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 551 | 552 | 1103
Education [Count of Participants; unit: Participants]
  Less than high school | 39 | 43 | 82
  High school | 174 | 188 | 362
  Some college | 182 | 156 | 338
  Bachelor's degree or higher | 156 | 165 | 321
Income [Count of Participants; unit: Participants]
  Less than $25,000 | 141 | 132 | 273
  $25,000 - $49,999 | 160 | 148 | 308
  $50,000 - $74,999 | 111 | 111 | 222
  $75,000 and above | 139 | 161 | 300
Years of diagnosis [Mean (Standard Deviation); unit: years] | 11.47 (8.26) | 11.24 (7.81) | 11.35 (8.03)
Self-reported health [Count of Participants; unit: Participants]
  Excellent | 27 | 33 | 60
  Very good | 158 | 158 | 316
  Good | 233 | 232 | 465
  Fair | 103 | 106 | 209
  Poor | 30 | 23 | 53
No. of hypoglycemic events in the past 6 months [Count of Participants; unit: Participants]
  None | 278 | 293 | 571
  1 time | 80 | 80 | 160
  2-5 times | 144 | 134 | 278
  More than 5 times | 49 | 45 | 94
No. of HbA1c level measured in past 6 months [Count of Participants; unit: Participants]
  None | 31 | 41 | 72
  1 time | 253 | 239 | 492
  More than 2 times | 246 | 261 | 507
  Don't know | 21 | 11 | 32
Most recent HbA1c level [Count of Participants; unit: Participants]
  Over 9.0% | 37 | 21 | 58
  Over 8.0% but under 9.0% | 46 | 59 | 105
  Over 7.0% but under 8.0% | 144 | 153 | 297
  Under 7.0% | 232 | 228 | 460
  Don't know | 92 | 91 | 183
Type of diabetes medicine used [Count of Participants; unit: Participants]
  No prescription medicine | 62 | 37 | 99
  Only pills | 321 | 345 | 666
  Only injections/shots | 48 | 42 | 90
  Pills and injections/shots | 119 | 127 | 246
  Refused | 1 | 1 | 2
Complications [Count of Participants; unit: Participants]
  Yes | 237 | 226 | 463
  No | 314 | 326 | 640
Other chronic conditions [Count of Participants; unit: Participants]
  Yes | 461 | 460 | 921
  No | 90 | 92 | 182

OUTCOME MEASURES:

1. Primary Outcome: Patient Medication Preference as Estimated by a Choice Model
Description: Preference estimate for each medicine attribute level from a conditional logit regression analysis. For each arm, there were six attributes of the medication, with 3 levels each. Within each attribute the parameter estimates for each of the levels sum to 0. If a parameter estimate for a level is above (below) 0 then the parameter is higher (lower) than average for that medication attribute.
Time Frame: One-time survey
Population: Respondents who completed the survey.
Measure: Mean (95% Confidence Interval); unit: utility of
Groups:
- Best-Worst Scaling (Case 2): Preference measured by best-worst scaling (case 2) survey method
  Best-Worst Scaling (Case 2): Respondents receive questions asking them to choose the best and worst features of a hypothetical medication.
Arm/Group | Best-Worst Scaling (Case 2) | Discrete Choice Experiment
Number analyzed (Participants) | 551 | 552
utility of
  HbA1c decrease by 1% | 0.983 [0.903 to 1.064] | 0.362 [0.254 to 0.470]
  HbA1c decrease by 0.5% | 0.284 [0.180 to 0.387] | 0.261 [0.165 to 0.358]
  HbA1c decrease by 0% | -1.267 [-1.369 to -1.165] | -0.623 [-0.724 to -0.522]
  HbA1c stable 6 days/week | 0.859 [0.789 to 0.928] | 0.395 [0.303 to 0.488]
  HbA1c stable 4 days/week | -0.030 [-0.106 to 0.046] | 0.073 [-0.027 to 0.174]
  HbA1c stable 2 days/week | -0.828 [-0.894 to -0.762] | -0.469 [-0.564 to -0.373]
  No hypoglycemia | 0.640 [0.562 to 0.718] | 0.325 [0.243 to 0.406]
  Hypoglycemia during the day | -0.145 [-0.224 to -0.065] | 0.104 [0.016 to 0.193]
  Hypoglycemia during day and/or night | -0.495 [-0.562 to -0.428] | -0.429 [-0.510 to -0.348]
  No nausea | 1.158 [1.075 to 1.240] | 0.739 [0.629 to 0.849]
  Nausea for 30 min/day | -0.262 [-0.345 to -0.179] | 0.236 [0.162 to 0.310]
  Nausea for 90 min/day | -0.896 [-0.961 to -0.830] | -0.975 [-1.084 to -0.866]
  1 pill/day | 0.561 [0.504 to 0.618] | 0.456 [0.353 to 0.560]
  2 pills/day | 0.128 [0.054 to 0.202] | 0.348 [0.230 to 0.467]
  1 pill and 1 injection/day | -0.689 [-0.763 to -0.614] | -0.805 [-0.911 to -0.699]
  $10 out-of-pocket cost | 0.900 [0.821 to 0.980] | 0.550 [0.405 to 0.696]
  $30 out-of-pocket cost | -0.051 [-0.134 to 0.032] | 0.077 [-0.116 to 0.271]
  $50 out-of-pocket cost | -0.850 [-0.919 to -0.780] | -0.628 [-0.791 to -0.464]

2. Primary Outcome: Weight Respondents Assign to Medication Attribute (Relative Attribute Importance) Assessed by a Choice Model
Description: Relative attribute importance (RAI) for each attribute in each arm measures the overall importance of that attribute. It is estimated by subtracting the lowest parameter estimate from the highest parameter estimate within each attribute. The RAI was then re-scaled on a 0 to 10 scale with 0 demonstrating no importance and 10 reflecting the most important attribute in each arm.
Time Frame: One-time survey
Population: Respondents who completed the survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Best-Worst Scaling (Case 2) | Discrete Choice Experiment
Number analyzed (Participants) | 551 | 552
units on a scale
  HbA1c decrease | 10 [9.540 to 10.460] | 5.745 [5.182 to 6.308]
  Duration of stable HbA1c | 7.496 [7.159 to 7.833] | 5.040 [4.453 to 5.626]
  Frequency of hypoglycemia | 5.043 [4.689 to 5.398] | 4.395 [3.878 to 4.912]
  Duration of nausea | 9.125 [8.755 to 9.494] | 10 [9.567 to 10.433]
  Treatment burden | 5.553 [5.225 to 5.880] | 7.358 [6.668 to 8.048]
  Out-of-pocket cost | 7.777 [7.406 to 8.147] | 6.873 [5.745 to 8.001]

3. Secondary Outcome: Self-reported Difficulty in Understanding and Answering the Survey Questions
Description: Questions that asked the respondents to evaluate if the Best-Worst Scaling (BWS) or Discrete Choice Experiment (DCE tasks were easy to understand and answer.
Time Frame: One-time survey
Population: Respondents who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Best-Worst Scaling (Case 2) | Discrete Choice Experiment
Number analyzed (Participants) | 551 | 552
Participants
  I found it easy to understand the questions: Strongly disagree | 20 | 13
  I found it easy to understand the questions: Disagree | 49 | 36
  I found it easy to understand the questions: Neither agree nor disagree | 123 | 111
  I found it easy to understand the questions: Agree | 248 | 292
  I found it easy to understand the questions: Strongly agree | 105 | 99
  I found it easy to understand the questions: Refused | 6 | 1
  I found it easy to answer all the questions: Strongly disagree | 18 | 15
  I found it easy to answer all the questions: Disagree | 73 | 61
  I found it easy to answer all the questions: Neither agree nor disagree | 133 | 123
  I found it easy to answer all the questions: Agree | 225 | 262
  I found it easy to answer all the questions: Strongly agree | 94 | 89
  I found it easy to answer all the questions: Refused | 8 | 2
  My answers are consistent with my preferences: Strongly disagree | 8 | 12
  My answers are consistent with my preferences: Disagree | 9 | 13
  My answers are consistent with my preferences: Neither agree nor disagree | 82 | 83
  My answers are consistent with my preferences: Agree | 314 | 318
  My answers are consistent with my preferences: Strongly agree | 132 | 126
  My answers are consistent with my preferences: Refused | 6 | 0

ADVERSE EVENTS:
Description: Adverse events were not collected
Arm/Group | Best-Worst Scaling (Case 2) | Discrete Choice Experiment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No